CLINICAL TRIAL: NCT07211841
Title: Correlative Analysis Between Magnetic Resonance Spectroscopy (MRS) and Essential Clinicobiological Data in Glioblatoma Multiforme (GBM)
Acronym: GLIOMIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0123
Record Dates: First submitted 2025-09-04; First posted 2025-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma; MRI Spectroscopy; Tumor Microenvironment; Biomarkers / Blood
Keywords: Glioblastoma; MRI spectroscopy; Tumor microenvironment; biomarkers
MeSH Terms: conditions — Glioblastoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRS study — Thirty patients newly diagnosed with GBM will be included in this study. The study will be conducted without any major modification of the standard management of GBM.
  The MRS study will be performed at the time of the initial MRI examination (morphological MRI sequences performed on 3T Philipps). The MRS will be performed on the most agressive part of the tumor : monovoxel PRESS MRS sequence with 3 echo times : 35, 144 and 288 ms. Spectra processing with Philipps software returns relative quantifications > 7 ratios (choline/creatin, Glucose/creatin, glutamine/creatin, N-Acetyl aspartate/creatin, myoinositol/creatin, phsopholipids/creatin, lactate/creatin, acetate/creatin). With this experimental design, the additional time required for MRS acquisition is 10 min /patient.
Biological: blood samples — Routine basic clinical and biological analyses will be collected during the project. In addition, 2 blood samples (5 mL each time) will be obtained at the time of inclusion (pre-therapeutic) and one month after completion of the initial therapeutic cycle (surgery + radiochemotherapy). The plasma samples will be used to measure fibrinogen, lactate and choline concentrations. In addition, a metabolomic study of plasma will be performed w

SUMMARY:
Glioblastoma multiforme (GBM) is the most common primary brain tumor, and it is well-known to be associated with a poor prognosis. MRI is the key medical technique for the diagnosis and the follow-up of GBM. By allowing for MRS studies, MRI permits a non-invasive characterization of the TME of GBM, including their metabolic characterization. The investigators propose to address the link between the MRS profile of GBM and basic clinical and biological parameters, with the aim of : i) identifying correlations between these parameters, ii) attempting to integrate clinical, biological and spectroscopic profiles of GBM. The investigators plan to recruit 30 newly diagnosed GBM patients for which surgery / radiochemotherapy will be proposed in the Medical oncology unit of Amiens University Hospital. Following inclusion of patients with probable GBM, MRS study will be performed during the first (pre-therapeutic) MRI examination. Basic clinical and biological parameters of the blood (CRP, complete blood count, fibrinogen, lactate and choline) will be assessed. A metabolomic study will also be performed on the plasma of GBM patients before any therapeutics. A second biological, post-therapeutic assesment (one month after surgery/radiochemotherapy) will allow the same analyses (basic biological parameters + plasma metabolomics), in order to examine the stability of the blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively identified in the multidisciplinary consultation meeting of neurooncology with a new diagnosis of GBM / a probable diagnosis of GBM. - Patients that have not started radiochemotherapy ;
* Adult > 18 yrs
* socially-insured,
* having given consent.

Exclusion Criteria:

* minor patients,
* pregnant/lactating women,
* patients under guardianship,
* curatorship,
* protection of justice or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Correlations between initial spectroscopic parameters, basic clinical and biological informations | 12 months
  correlations between initial spectroscopic parameters of the tumor, basic clinical information and biological assessment of the blood in a cohort of newly-diagnosed GBM
  Blood parameters are choline, creatinine, lactate, glutamate/glutamine, alanine, glycine. For each parameter, absolute concentrations will be measured. A Z transformation will be used as a preliminary step ahead of all analyses (heat map construction, testing correlations).

SECONDARY OUTCOMES:
Variation from baseline of blood parameters | at 1 month
  Variation from baseline of blood parameters at one month after surgery/radiochemotherapy in each patient. Blood parameters are choline, creatinine, lactate, glutamate/glutamine, alanine, glycine. For each parameter, absolute concentrations will be measured. A Z transformation will be used as a preliminary step ahead of all analyses (heat map construction, testing correlations).
Progression-free survival | at 12 months
Overall survival | at 12 months
Correlation of biological and metabolomic data with progression-free survival | at 12 months
  Blood parameters are choline, creatinine, lactate, glutamate/glutamine, alanine, glycine. For each parameter, absolute concentrations will be measured. A Z transformation will be used as a preliminary step ahead of all analyses (heat map construction, testing correlations).
Correlation of biological and metabolomic data with overall survival | at 12 months
  Blood parameters are choline, creatinine, lactate, glutamate/glutamine, alanine, glycine. For each parameter, absolute concentrations will be measured. A Z transformation will be used as a preliminary step ahead of all analyses (heat map construction, testing correlations).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No